CLINICAL TRIAL: NCT05033145
Title: Evaluation of the Safety and Clinical Efficacy of AZVUDINE: Randomized, Double-blind, Placebo-controlled Study in Mild Stage Patients Infected With the SARS-CoV-2 Virus
Brief Title: Study on Safety and Clinical Efficacy of AZVUDINE in Initial Stage COVID-19 Patients (SARS-CoV-2 Infected)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HRH Pharmaceuticals Limited (Other)
Collaborators: GALZU INSTITUTE OF RESEARCH, TEACHING, SCIENCE AND APPLIED TECHNOLOGY, Brazil (Unknown); Clinical Research Unit / High Complexity Center (CRU/HCC) / Galzu Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FNC IGZ-2
Record Dates: First submitted 2020-12-04; First posted 2021-09-02 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2021-09

CONDITIONS: COVID-19
Keywords: AZVUDINE; SARS-CoV-2; COVID-19; FNC
MeSH Terms: conditions — COVID-19 | interventions — azvudine; Cytosine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, parallel, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZVUDINE (Experimental): Experimental:
  AZVUDINE 1mg tablet
  Interventions:
  AZVUDINE 1mg tablet, 5 tablets QD + standard treatment, for up to 14 days
  Interventions: Drug: AZVUDINE
- AZVUDINE placebo (Placebo Comparator): Control:
  AZVUDINE placebo
  Intervention:
  AZVUDINE placebo tablet, 5 tablets QD + standard treatment, for up to 14 days
  Interventions: Drug: AZVUDINE placebo

INTERVENTIONS:
Drug: AZVUDINE — AZVUDINE 5 tablets QD + standard treatment, for up to 14 days
  Other Names: AZVUDINE 1 mg tablets; FNC; 4-amino-1-((2R,3S,4R,5R)-5-azido-3-fluoro-4-hydroxy-5-(hydroxymethyl)tetrahydrofuran-2-yl)pyrimidine-2(1H)-one; 1-(4-Azido-2-deoxy-2-fluoro-beta-D- arabino Ribo-furanosyl) cytosine, FNC
  Arms: AZVUDINE
Drug: AZVUDINE placebo — 5 tablets QD + standard treatment, for up to 14 days
  Other Names: Placebo
  Arms: AZVUDINE placebo

SUMMARY:
Phase III, single-center with co-participating units, randomized, double-blind, parallel, placebo-controlled clinical study

DETAILED DESCRIPTION:
Hypothesis:

AZVUDINE has a therapeutic potential and safety profile for the treatment of patients infected with SARS-CoV-2.

Goals:

Main goal:

To evaluate the efficacy and safety of AZVUDINE (FNC) in patients infected with SARS-COV-2, in a mild stage;

Specific objective:

To assess the clinical outcome of mild-stage SARS-CoV-2 infected participants treated with AZVUDINE (FNC) versus placebo

Statistical planning:

Statistical description: all statistical tests are performed by bilateral testing. A significance level of 5% will be adopted.

Baseline analysis: including subject distribution, data demographics, and baseline analysis.

ELIGIBILITY:
Inclusion Criteria:

Individuals who present the following characteristics will be included in this study:

1. Age ≥18 years, regardless of gender;
2. Fluorescence RT-PCR test result of respiratory or blood samples must be positive for COVID-19, or viral gene sequencing of respiratory tract samples must be highly homologous to COVID-19; Individuals with COVID-19 must meet the diagnostic criteria in the "latest version of clinical guidelines for COVID-19" issued by the World Health Organization (WHO) on June 4, 2020;
3. Symptomatic patients who meet the case definition for COVID-19, according to WHO, without evidence of bacterial pneumonia or hypoxia (Sat O2 < 95%) P. [score 1-3];
4. Voluntary participation and signing of the informed consent form.

Exclusion Criteria:

Individuals who present one or more of the following characteristics will not be eligible to participate in this study:

1. Know or suspect that you are allergic to any of the components of AZVUDINE tablets (inactive ingredients: microcrystalline cellulose, lactose hydrate, polyvinylpyrrolidone K30, croscarmellose sodium, magnesium stearate);
2. Individual presenting shortness of breath and Sat O2 < 95%; or any other symptom requiring treatment through hospital admission;
3. Patients with liver disease (total bilirubin ≥2mg/dL, ALT/TGP e AST/TGO ≥5 times above normal limit);
4. Pactients with a history of known liver disease (cirrhosis with ChildPugh classification B and C);
5. Patients with a history of renal insufficiency (glomerular filtration rate < 60mL/min/1,73m2);
6. Patients with history of congestive heart failure (NYHA ¾ grade), untreated symptomatic arrhythmias ormyocardial infarction within 6 months;
7. Individuals with malabsorption syndrome, or other conditions affecting gastrointestinal absorption, and circumstances in which patients require intravenous nutrition, or cannot take medications orally or nasogastrically;
8. Total neutrophil count <750 cells/L;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Proportion of patients hospitalized during the study through day 28 | Day 14 to Day 30
  WHO clinical progression ordinal scale (Jun/2020), Score 4 to 10.Health Organization Ordinal Clinical Progression Scale (WHO, Jun/2020; scale 0 [asymptomatic] to 10 [death]), with score 4 to 7.
Proportion of participants with a clinical outcome of CURE during the study; | Day 14 to Day 30
  The clinical outcome of cure is defined in this protocol as the absence of viral RNA in samples collected and clinical conditions for outpatient discharge.

SECONDARY OUTCOMES:
Improvement in clinical status in at least one category compared to screening | Day 14 to Day 30
  Ordinal Scale of Clinical Improvement (WHO, Jun/2020)
Severity and duration of symptoms: fever, cough, fatigue or tiredness, breathlessness, myalgia, nasal congestion or runny nose, sore throat, headache, chills, nausea, vomiting, anosmia, ageusia. | Day 1 to Day 14
  Intensity (1= Mild; 2= Moderate; 3= Severe; 4= Critical)
Changes in kidney function | Day 1 to Day 30
  Change in urea/creatinine
Changes in liver function | Day 1 to Day 30
  Changes in ALT/AST
Time of use of AZVUDINE until the second negative conversion of RT-PCR | Day 1 to Day 14
  Rate of change in biochemical markers of inflammatory function in relation to the physiological reference intervals between the AZVUDINA and PLACEBO groups.
Evaluation of SARS-CoV-2 viral load negative conversion time by RT-PCR between AZVUDINE group (FNC) and control group | Day 1 to Day 28
  RT-PCR performed on treatment days.
Occurrence of drug interactions | Day 1 to Day 14
  Monitoring of concomitant medication
Assessment of liver function biochemical markers (AST/TGO, ALT/TGP, ALP, GGT, BIL total, and direct BIL) | Day 1 to Day 60
  Rate of change in biochemical markers of hepatic function in relation to the physiological reference intervals between the AZVUDINA and PLACEBO groups.
All-cause mortality rate during the study | Day 1 to Day 60
  mortality and its causes
Frequency and intensity of adverse events, unexpected adverse events, and serious adverse events | Day 1 to Day 30
  Intensity of adverse events (1= Mild; 2= Moderate; 3= Severe; 4= Critical)
Proportion of comorbidity-related worsening [Obesity, diabetes, alcoholism, smoking, lung disease] | Day 1 to Day 30
  relationship between comorbidities and aggravations
hospitalization for all causes occurring in post-treatment period | Day 1 to Day 60
  hospitalization for all causes after treatment
To assess the tolerability of using AZVUDINE (FNC) at 5mg/day | Day 1 to Day 14
  calculation of participants who completed treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sheila P Figueiredo, Nurse,MSc, Study Chair — Galzu Institute
Locations (7):
- Brazil (7):
  - Hospital Moacyr Gomes de Azevedo, Cambuci, Rio de Janeiro
  - Clinical Research Unit / High Complexity Center (CRU/HCC) / Galzu Institute, Campos dos Goytacazes, Rio de Janeiro
  - Hospital Santa Casa de Misericórdia de Campos, Campos dos Goytacazes, Rio de Janeiro
  - Unidade de Pesquisa Clínica / Centro de Alta Complexidade, Campos dos Goytacazes, Rio de Janeiro
  - Unidade Pré Hospitalar São José, Campos dos Goytacazes, Rio de Janeiro
  - Hospital de Itaocara, Itaocara, Rio de Janeiro
  - Hospital Armando Vidal, São Fidelis, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] da Silva RM, Gebe Abreu Cabral P, de Souza SB, Arruda RF, Cabral SPF, de Assis ALEM, Martins YPM, Tavares CAA, Viana Junior AB, Chang J, Lei P. Serial viral load analysis by DDPCR to evaluate FNC efficacy and safety in the treatment of mild cases of COVID-19. Front Med (Lausanne). 2023 Mar 14;10:1143485. doi: 10.3389/fmed.2023.1143485. eCollection 2023. PMID 37007788